CLINICAL TRIAL: NCT00313924
Title: The Applicability of the OAB Assessment Tool for Evaluation of Treatment Efficacy of Overactive Bladder.
Brief Title: Assessing the OAB-8 Questionnaire as a Tool to Measure Treatment Outcome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: oab.CTIL
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Overactive Bladder
Keywords: URGENCY FREQUENCY SYNDROME; URGE INCONTINENCE
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: DETRUSITOL

SUMMARY:
OAB is a widespread medical problem affecting 6- 30% of the population (both sexes and all age groups) in Europe1 and 16%2-18%3 of the US and Canadian population. Nevertheless only a small proportion of this group turns to seek medical help. Once treated, evaluation of treatment outcome is problematic since outcome measures for success vary widely (i.e. improvement in number of incontinence episodes, number of urge episodes, change in frequency and nocturia etc) but do not include measures of patient reported outcomes.

The OAB Assessment Tool is a self-administered questionnaire (8-question self-filled survey) primarily intended to identify patients with symptoms of OAB. The same comparable information could be obtained after a certain treatment period, thus providing accurate and precise measures of success. It could also offer insight to the changes of the different parameters that make up the problem. Due to its ease of administration and its high specificity in assessing OAB, the OAB Assessment Tool seems to be optimal for this objective.

DETAILED DESCRIPTION:
This study will be a non-randomised, non-placebo controlled prospective clinical trial.

We intend to recruit approximately 100 patients that will receive and fill out the questionnaire before and after medical treatment with detrusitol 4mg.

Study protocol will receive approval of the local ethical committee.

Method:

Twenty general practitioners (GP) will actively participate in the recruitment and treatment of these patients. After a brief inquiry, patients with urinary complaints will be offered the option of completing the OAB-V8 questionnaire and to participate in this trial if eligible.

After the patient fills out the OAB-V8 and is found fit for this study, the patient will receive accurate information regarding the study and will sign an informed consent form.

Protocol:

The study will consist of 2 visits, visit 1 pre and visit 2 post-treatment with Detrusitol 4mg.

Visit I:

Randomly selected patients will be requested to complete the OAB -V8 questionnaire. Those with a score >8 points will be eligible for inclusion. They will complete an informed consent form and will undergo a basic medical history. Patients will then be given treatment with detrusitol 4mg once daily (a total of 28 tablets). They will also be required to fill out a voiding/frequency and urgency chart for three days prior to commencing treatment and again three days before finishing the treatment period (day 25 of the treatment period) to confirm diagnosis of OAB. Patients will also be asked questions and lab work will be performed to rule out patients with other Urinary Conditions.

Information on side effects and a contact number 24/7 for any question or problem that arises will be provided. After the end of one-month treatment, patients will return for their 2nd and final visit.

Twenty-eight tablets of Detrusitol 4mg will be provided to every patient. Visit II: Patients will be evaluated with regard to effect of treatment by completing the OAB-V8 questionnaire again. On this visit, according to the physicians' professional consideration, satisfied patients will receive a prescription of Detrusitol 4mg for continuing treatment.

The statistical methods that will be employed will include Chi Square and Fisher exact tests, and logistic regression (the logistic will be run mainly for covariates such as age, gender and baseline symptom severity score to predict who achieve a 10 point change in symptom bother scale. Software utilised will include SAS and JMP.

ELIGIBILITY:
Inclusion Criteria:

1. OAB score of ≥ 8
2. Age 20-80 years old
3. Patients must comply and agree to the requirement of taking only Detrusitol 4mg and no other new medication affecting the lower urinary tract system

Exclusion criteria:

1. Patients that are on any other treatment (whether medical or conservative) for OAB.
2. Patients with documented UTI.
3. Patients who have demonstrated hypersensitivity to the drug or its ingredients.
4. Where Detrusitol is contraindicated (i.e. patients with severe outlet obstruction, gastric retention, or uncontrolled narrow-angle glaucoma).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-02; Study Completion 2006-03

PRIMARY OUTCOMES:
A significant correlation between reduced urinary symptoms and a reduction of more than 10 points in the OAB-8 score.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Healthcare Center, Haifa, Israel

REFERENCES:
- [Background] Corcos J, Schick E. Prevalence of overactive bladder and incontinence in Canada. Can J Urol. 2004 Jun;11(3):2278-84. PMID 15287994
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Milsom I, Stewart W, Thuroff J. The prevalence of overactive bladder. Am J Manag Care. 2000 Jul;6(11 Suppl):S565-73. PMID 11183899